CLINICAL TRIAL: NCT01334957
Title: A Multi-Center, Open-Label, Surgical Surveillance Trial To Evaluate The Safety And Efficacy Of A Shortened Infusion Time of Intravenous Ibuprofen
Brief Title: Surgical Surveillance Trial to Evaluate a Shortened Infusion Time of Intravenous Ibuprofen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPI-CL-016
Record Dates: First submitted 2011-04-12; First posted 2011-04-13 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravenous ibuprofen (Experimental): Intravenous ibuprofen (800 mg intravenous ibuprofen administered intravenously over 5-10 minutes) will be administered as a single dose during the 10 minute Treatment Period.
  Interventions: Drug: Intravenous ibuprofen

INTERVENTIONS:
Drug: Intravenous ibuprofen — 800 mg intravenous ibuprofen administered intravenously over 5-10 minutes
  Other Names: Caldolor

SUMMARY:
The primary objective of this study is to determine the safety of a single dose of intravenous ibuprofen administered over 5-10 minutes for the preemptive treatment of postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgery with anticipated need for postoperative analgesia

Exclusion Criteria:

1. Patients with inadequate IV access
2. Patients <18 years of age
3. History or allergy or hypersensitivity to any component of intravenous ibuprofen, aspirin (or aspirin related products) or non-steroidal anti-inflammatory drug (NSAIDs)
4. Active hemorrhage or clinically significant bleeding
5. Pregnant or nursing
6. Patients in the peri-operative period in the setting of coronary artery bypass graft (CABG) surgery
7. Inability to understand the requirements of the study, be willing to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]), and agree to abide by the study restrictions
8. Refusal to provide written authorization for use and disclosure of protected health information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Art P Wheeler, M.D., Study Director — Cumberland Pharmaceuticals, Inc.
Locations (22):
- United States (22):
  - UC San Diego Regional Center, La Jolla, California
  - Neurovations (Queen of the Valley Hospital), Napa, California
  - University of Miami Health System, Miami, Florida
  - Sheridan Clinical Research, Plantation, Florida
  - RUSH Univ. Medical Center, Chicago, Illinois
  - Univ. of Kansas Medical Center, Kansas City, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Detroit Medical Center, Detroit, Michigan
  - North Mississippi Sports Medicine & Orthopaedic Clinic, Tupelo, Mississippi
  - Albany Medical Center, Albany, New York
  - State of New York Downstate Medical Center (SUNY), Brooklyn, New York
  - North Shore - Long Island Jewish Health System, Manhasset, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Penn State College of Medicine, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Hendersonville Hospital/Comprehensive Pain Specialists, Hendersonville, Tennessee
  - Parkland Memorial, Dallas, Texas

REFERENCES:
- [Derived] Gan TJ, Candiotti K, Turan A, Buvanendran A, Philip BK, Viscusi ER, Soghomonyan S, Bergese SD; Intravenous Ibuprofen Surgical Surveillance Trial Investigational Sites. The shortened infusion time of intravenous ibuprofen, part 2: a multicenter, open-label, surgical surveillance trial to evaluate safety. Clin Ther. 2015 Feb 1;37(2):368-75. doi: 10.1016/j.clinthera.2014.12.006. Epub 2015 Jan 13. PMID 25592331

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult hospitalized patients undergoing surgery
Pre-assignment Details: Patients who met all the inclusion and none of the exclusion criteria during the Screening /Baseline Period were enrolled into the study.
  Subjects could not have a history of allergy or hypersensitivity to any component of intravenous ibuprofen, aspirin (or aspirin related products) or NSAIDS.
Groups:
- Intravenous Ibuprofen: Intravenous ibuprofen (800 mg intravenous ibuprofen administered intravenously over 5-10 minutes) will be administered as a single dose during the 10 minute Treatment Period. A minimum of one dose of intravenous ibuprofen will be administered. At the discretion of the investigator, up to three additional doses of 800 mg intravenous ibuprofen may be administered at six hour intervals.
  Intravenous ibuprofen: 800 mg intravenous ibuprofen administered intravenously over 5-10 minutes
Period: Overall Study
Arm/Group | Intravenous Ibuprofen
Started | 300
Received Single Dose | 252
Received Multiple Doses | 48
Completed | 300
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Formal sample size calculations were not performed. The intent is to enroll 300 patients to provide descriptive safety and efficacy data.
Arm/Group | Intravenous Ibuprofen
Number analyzed (Participants) | 300
Age, Customized [Number; unit: years] — Greater than or equal to 18 years of age
  years
    Greater than or equal to 18 years of age | 300
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189
  Male | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 271
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 60
  White | 229
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 300

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Safety of a Single Dose of Intravenous Ibuprofen Over 5-10 Minutes for the Reduction of Pain.
Description: The incidence of treatment-emergent serious adverse events occurring in the six hours following administration of the first dose of intravenous ibuprofen
Time Frame: 6 hours
Measure: Number; unit: Number of Serious Adverse Events
Arm/Group | Intravenous Ibuprofen
Number analyzed (Participants) | 252
Number of Serious Adverse Events | 8

2. Primary Outcome: To Determine the Safety of a Single Dose of Intravenous Ibuprofen Administered Over 5-10 Minutes for the Reduction of Post-operative Pain.
Description: The incidence of treatment-emergent adverse events occurring in the six hours following administration of the first dose of intravenous ibuprofen
Time Frame: 6 hours
Measure: Number; unit: Number of Adverse Events
Arm/Group | Intravenous Ibuprofen
Number analyzed (Participants) | 252
Number of Adverse Events | 49

3. Secondary Outcome: To Determine the Safety of a Multiple Doses of Intravenous Ibuprofen Over 5-10 Minutes for the Reduction of Pain.
Description: The incidence of treatment-emergent serious adverse events occurring in the six hours following administration of the last dose of intravenous ibuprofen
Time Frame: 6 hours
Measure: Number; unit: Number of Serious Adverse Events
Arm/Group | Intravenous Ibuprofen
Number analyzed (Participants) | 48
Number of Serious Adverse Events | 0

4. Secondary Outcome: To Determine the Safety of a Multiple Doses of Intravenous Ibuprofen Administered Over 5-10 Minutes for the Reduction of Post-operative Pain.
Description: The incidence of treatment-emergent adverse events occurring in the six hours following administration of the last dose of intravenous ibuprofen
Time Frame: 6 hours
Measure: Number; unit: Number of Adverse Events
Arm/Group | Intravenous Ibuprofen
Number analyzed (Participants) | 48
Number of Adverse Events | 16

5. Secondary Outcome: To Determine the Safety of a Multiple Doses of Intravenous Ibuprofen Administered Over 5-10 Minutes for the Reduction of Post-operative Pain.
Description: Visual Analog Scale (VAS) assessments following surgery. The VAS is a continuous scale compromised of a horizontal line, one hundred millimeters in length, anchored by 2 verbal descriptors (No Pain, Worst Possible Pain). The VAS is self-completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance, in mm, on the 100 mm line between the "No Pain" anchor and the subject's mark. The score would be between o and 100.
Time Frame: 6 hours
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intravenous Ibuprofen
Number analyzed (Participants) | 228
units on a scale | 30.9 [27.5 to 34.2]

ADVERSE EVENTS:
Time Frame: During and after dosing with intravenous ibuprofen until 6 hours following the last dose of intravenous ibuprofen
Arm/Group | Intravenous Ibuprofen
Serious Adverse Events (participants affected / at risk) | 8/300
Other Adverse Events (participants affected / at risk) | 49/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Ibuprofen (N=300)
Abdominal Compartment Syndrome (Gastrointestinal disorders) | 1 (1)
Peritoneal Adhesions (Gastrointestinal disorders) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1)
Airway Complication Of Anaesthesia (Injury, poisoning and procedural complications) | 1 (1)
Oxygen Saturation Decreased (Investigations) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Ibuprofen (N=300)
Infusion Site Pain (General disorders) | 34 (34)
Nausea (Gastrointestinal disorders) | 10 (10)
Flatulence (Gastrointestinal disorders) | 9 (9)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 10 (10)
Bradycardia (Cardiac disorders) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No